CLINICAL TRIAL: NCT05516433
Title: Effect of Imipenem and Meropenem on the Digestive Microbiota and the Emergence and Carriage of Multidrug-resistant Bacteria
Acronym: MERIMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MERIMI
Record Dates: First submitted 2022-08-17; First posted 2022-08-25 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Enterobacteriaceae Infections
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Imipenem: Prescribing rules differ from one department to another: Imipenem is the preferred drug at Saint-Joseph Hospital.
- Meropenem: Prescribing rules differ from one department to another: Meropenem is the preferred carbapenem at Avicenne Hospital.

SUMMARY:
Among enterobacteria, ESBL production is the leading cause of multidrug resistance. The first cases of ESBL-producing Enterobacteriaceae (EBLSE) infections were described in the 1980s and subsequently spread worldwide.

Since the turn of the century, the prevalence of EBLSE infections, particularly among E. coli and K. pneumoniae, has increased dramatically. The emergence of multidrug-resistant enteric bacteria (MRE) is currently a real public health problem. The European network for monitoring antibiotic resistance in cooperation with Santé Publique France evaluated the rate of resistance to third generation cephalosporins (C3G) among clinical strains at 10.2% for Escherichia coli and 28.8% for Klebsiella pneumoniae. The consequences of infections with multi-resistant enteric bacteria, mainly represented by ESBL, are currently well known, both from an individual point of view (increased mortality and length of hospitalization) and from a collective point of view (increased costs of care).

The current reference treatment for ESBL-producing Enterobacteriaceae infections is based on carbapenems.

Imipenem and meropenem are the two most commonly used carbapenems in clinical practice. Despite their similar spectrum of action, these two molecules have different pharmacokinetic properties, notably concerning their half-life and their elimination routes (mainly urinary for imipenem, mixed: biliary and urinary for meropenem).

Some studies have suggested that imipenem has a low impact on the digestive microbiota. However, no studies comparing the impact of imipenem and meropenem have been conducted.

Woerther et coll. explained in their work that the digestive microbiota confers resistance to colonization by MREs. The impact of antibiotics on the microbiota probably leads to a breakdown of this barrier and a loss of this resistance to colonization. Moreover, each antibiotic therapy does not impact the digestive microbiota in the same way and it seems that antibiotics with a high activity against strict anaerobic species and/or a high biliary elimination are the most impacting. It is therefore essential, in the era of multidrug resistance, to look at the influence of antibiotics on the digestive microbiota and on the emergence and carriage of MRE.

In a context where the incidence of multi-resistant bacteria is constantly increasing, it seems relevant to conduct a study aiming at comparing the respective impact of the use of imipenem and meropenem on the emergence of MRE and on the digestive microbiota at the individual level. This study aims at comparing the microbiological impact (in terms of emergence of bacterial resistance and in terms of impact on the diversity of cultivable digestive bacteria). It will be a comparative study with matching of patients according to age, service and previous duration of hospitalization. Indeed, the usual management of patients with an infection requiring treatment with a carbapenem is different between the 2 participating centers. Thus, according to the usual management of patients in these 2 participating centers, patients at Avicenne Hospital are treated with meropenem and patients at the Paris Saint-Joseph Hospital Group with imipenem, except in the case of a need for a high daily dose (osteoarticular infection, for example) due to the neurological toxicity of imipenem at high dosage. In the case of high-dose use, meropenem will be the preferred molecule.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient hospitalized in the intensive care unit of the Groupe Hospitalier Paris Saint-Joseph or the Avicenne Hospital
* Patient with an infection requiring probabilistic or documented treatment with a carbapenem (imipenem or meropenem)
* French speaking patient
* Patient or relative able to give his or her non-objection

Exclusion Criteria:

* Patients with a carbapenem allergy
* Pregnant or breastfeeding woman
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in the intensive care unit of the Groupe Hospitalier Paris Saint-Joseph or the Avicenne Hospital, with an infection requiring probabilistic or documented treatment with a carbapenem (imipenem or meropenem)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-01-22 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ecological impact of imipenem and meropenem on the microbiota (modification of bacterial diversity) | Month 1
  This outcome corresponds to the rate of modification in bacterial diversity judged by the loss of at least one bacterial species in the microbiota after initiation of antibiotic therapy.
Ecological impact of imipenem and meropenem on the microbiota (abundance) | Month 1
  This outcome corresponds to the rate of diminution in bacterial abundance within the microbiota, defined as a decrease of at least 2 logs in abundance.

SECONDARY OUTCOMES:
Evaluate the change in bacterial diversity | Month 1
  This outcome corresponds to the rate of loss of at least one bacterial species in the microbiota after initiation of antibiotic therapy.
Change in bacterial abundance | Month 1
  This outcome corresponds to the rate of loos corresponding to at least 2 log decrease in bacterial abundance.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PILMIS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Hôpital Avicenne, Bobigny
  - Groupe Hospitalier Paris Saint-Joseph, Paris

REFERENCES:
- [Background] Schwaber MJ, Navon-Venezia S, Kaye KS, Ben-Ami R, Schwartz D, Carmeli Y. Clinical and economic impact of bacteremia with extended- spectrum-beta-lactamase-producing Enterobacteriaceae. Antimicrob Agents Chemother. 2006 Apr;50(4):1257-62. doi: 10.1128/AAC.50.4.1257-1262.2006. PMID 16569837
- [Background] Gudiol C, Calatayud L, Garcia-Vidal C, Lora-Tamayo J, Cisnal M, Duarte R, Arnan M, Marin M, Carratala J, Gudiol F. Bacteraemia due to extended-spectrum beta-lactamase-producing Escherichia coli (ESBL-EC) in cancer patients: clinical features, risk factors, molecular epidemiology and outcome. J Antimicrob Chemother. 2010 Feb;65(2):333-41. doi: 10.1093/jac/dkp411. Epub 2009 Dec 3. PMID 19959544
- [Background] Woerther PL, Lepeule R, Burdet C, Decousser JW, Ruppe E, Barbier F. Carbapenems and alternative beta-lactams for the treatment of infections due to extended-spectrum beta-lactamase-producing Enterobacteriaceae: What impact on intestinal colonisation resistance? Int J Antimicrob Agents. 2018 Dec;52(6):762-770. doi: 10.1016/j.ijantimicag.2018.08.026. Epub 2018 Aug 31. PMID 30176355
- [Background] Ruppe E, Burdet C, Grall N, de Lastours V, Lescure FX, Andremont A, Armand-Lefevre L. Impact of antibiotics on the intestinal microbiota needs to be re-defined to optimize antibiotic usage. Clin Microbiol Infect. 2018 Jan;24(1):3-5. doi: 10.1016/j.cmi.2017.09.017. Epub 2017 Sep 29. No abstract available. PMID 28970162
- [Background] Ruppe E, Lixandru B, Cojocaru R, Buke C, Paramythiotou E, Angebault C, Visseaux C, Djuikoue I, Erdem E, Burduniuc O, El Mniai A, Marcel C, Perrier M, Kesteman T, Clermont O, Denamur E, Armand-Lefevre L, Andremont A. Relative fecal abundance of extended-spectrum-beta-lactamase-producing Escherichia coli strains and their occurrence in urinary tract infections in women. Antimicrob Agents Chemother. 2013 Sep;57(9):4512-7. doi: 10.1128/AAC.00238-13. Epub 2013 Jul 8. PMID 23836184